CLINICAL TRIAL: NCT01123746
Title: Utility of Laboratory Testing for Children With Seizure in Emergency Department
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Chou Hsiao-Feng, Department of Pediatrics, Taipei Medical University WanFang Hospital
Other Study IDs: 98088
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Seizure
Keywords: Seizure; electrolyte; risk factor
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: To evaluate the predisposing factors associated with abnormal laboratory findings in patients who came to the emergency room due to a first seizure.

Methods: Patients were divided into separate groups based on normal and abnormal laboratory results for sodium, potassium, calcium, and glucose. The difference in age, gender, whether this was the first attack, whether there was fever, whether there were gastrointestinal symptoms, the duration and pattern of the seizure, and whether there was a seizure at the emergency department, were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age: less than 18 years old
* The patient came to emergency department due to seizure
* The patient received blood sampling including serum sodium, potassium, calcium and glucose.

Exclusion Criteria:

* The patient came to the outpatient department.
* The patient did not received blood sampling at emergency room.
* The seizure occurred after admission.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 500 patients who come to wanfang hospital due to seizure
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Feng Chou, M.D., Principal Investigator — Pediatrics department, Wanfang hospital
Locations (1):
- Taipei Medical University-WanFang Hospital, Taipei, Taipei, Taiwan